CLINICAL TRIAL: NCT04339140
Title: A Phase 2 Study of Zafirlukast for the Treatment of Tumor-marker Only Relapsed Ovarian Cancer
Brief Title: Zafirlukast in Treatment of Marker Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Rushad Patell, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-814; 1R21CA231000-01A1 (NIH)
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Relapsed Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — zafirlukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zafirlukast (Experimental): Zafirlukast will be taken orally at a pre-determined dose 2x daily for 28 day cycle up to 1 year.
  Interventions: Drug: Zafirlukast

INTERVENTIONS:
Drug: Zafirlukast — Oral tablets, 2x daily for 28 day cycle up to 1 year
  Other Names: Accolate

SUMMARY:
This research study is evaluating the effectiveness of Zafirlukast to prevent tumor activity in participants with tumor marker-only relapsed ovarian cancer.

* The name of the study drug involved in this study is:
* Zafirlukast

DETAILED DESCRIPTION:
This is a single-arm Simon two-stage phase 2 clinical trial to determine whether zafirlukast reduces the tumor marker CA-125 as well the tendency to form blood clots in tumor marker-only relapsed ovarian cancer.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

* The name of the study drug involved in this study is:
* Zafirlukast

Eligible participants will receive study treatment for up to 1 year and will be followed for up to one year following treatment.

It is expected that about 30 people will take part in this research study.

The U.S. Food and Drug Administration (FDA) has not approved zafirlukast for this specific disease but it has been approved for other uses.

Zafirlukast is currently approved to be used for the treatment of asthma. It has been recently learned that Zakfirlukast demonstrates anti-tumor activity in laboratory studies of ovarian cancer. This means that these results were not found in humans.

The National Institutes of Health are supporting this research study by providing funding

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal cancer.
* Participants must have completed at least first-line platinum based chemotherapy and surgery with a response, in the opinion of the investigator, defined as no evidence of disease progression or rising CA-125 at any time during front-line treatment.
* Participants must meet criteria for tumor marker-only relapse, defined as CA-125 more than twice the upper limit of normal (35 U/mL) in the setting of a normal baseline CA-125 levels or CA-125 greater than twice the nadir count on two successive measurements for CA-125 values that remain above baseline without measurable radiographic disease.
* Minimum age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of zafirlukast in participants under 18 years of age with ovarian cancer, children are excluded from this study but will be eligible for future pediatric trials.
* Life expectancy of greater than 4 months.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%, see Appendix A).
* Participants must be able to swallow tablets.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,000/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤ 1.3 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2 × institutional ULN
  * Creatinine ≤ institutional ULN OR
  * Glomerular filtration rate (GFR) ≥45 mL/min/1.73 m2
* The effects of zafirlukast on the developing human fetus are incompletely characterized. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men are not eligible for this study.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Non-epithelial tumors (pure sarcomas) or ovarian tumors with low malignant potential (ie borderline tumors) or mucinous tumors. Mixed mullerian tumors or carcinosarcomas are allowed.
* Participants who have had cytotoxic chemotherapy including bevacizumab or radiotherapy within 4 weeks prior to entering the study. This does not include maintenance therapy (>8 weeks prior to enrollment of stable dose) with a PARP inhibitor, such as olaparib or niraparib. (PARP inhibitor, rucaparib is not allowed to be co-administered with CYP2C9 substrates as maintenance therapy as it could increase exposure to zafirlukast).
* Participants who have ongoing adverse effects from prior anti-cancer therapy greater than National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, v5.0) Grade 1, with the exception of Grade 2 non-hematologic toxicity such as alopecia and peripheral neuropathy.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to zafirlukast.
* Currently receiving anticoagulant therapy.
* Current daily use of aspirin (> 81 mg daily), clopidogrel (Plavix), cilostazol (Pletal), aspirin-dipyridamole (Aggrenox) (within 10 days) or considered to use regular use of higher doses of non-steroidal anti-inflammatory agents as determined by the treating physician (e.g. ibuprofen > 800 mg daily or equivalent).
* Participants receiving any medications or substances that are inhibitors or inducers of CYP2C9 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because zafirlukast is a class B agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with zafirlukast, breastfeeding should be discontinued if the mother is treated with zafirlukast.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rushad Patell, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single-arm study. All participants received 40 mg of Zafirlukast twice daily.
Period: Overall Study
Arm/Group | Zafirlukast
Started | 5
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zafirlukast
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: CA-125 Response Rate
Description: Response will be defined according to GCIG criteria which requires a reduction of CA-125 of > 50% relative to pre-treatment CA-125 level, maintained for at least 28 days
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | Zafirlukast
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: CTCAE v. 5
Arm/Group | Zafirlukast
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zafirlukast (N=4)
Headache (General disorders) | 1 (1) — Potentially related ot zafirlukast
Abdominal Pain (General disorders) | 3 (3) — Grade 1, not related to zafirlukast
Hypertension (Blood and lymphatic system disorders) | 1 (1) — Grade 2, unrelated to zafirlukast
Abdominal Bloating (General disorders) | 1 (1) — Grade 2, unrelated to zafirlukast

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT04339140/Prot_SAP_000.pdf